CLINICAL TRIAL: NCT00529204
Title: Effects Of Exenatide (Byetta®) On Liver Biochemistry, Liver Histology And Lipid Metabolism In Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: Effects Of Exenatide On Liver Biochemistry, Liver Histology And Lipid Metabolism In Patients With Fatty Liver Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of California, Davis (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200715325; H80-MC-X006 (Other: UC Davis)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Complications; Fatty Liver
Keywords: Fatty Liver; Nonalcoholic fatty liver disease; NAFDL; Diabetes; ALT; exenatide
MeSH Terms: conditions — Diabetes Complications; Fatty Liver; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exenatide (Experimental): exenatide 5 µg BID s.c. daily for 28 days, followed by 10 µg BID s.c. daily from day 29 to week 24
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — Subjects meeting the inclusion criteria will be treated with exenatide 5 µg BID s.c. for 3-7 days, followed by 10 µg BID s.c. daily to week 24
  Other Names: BYETTA

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH) are common complications of type 2 diabetes and leading causes of liver disease in the US and Europe. The prevalence of NAFLD and NASH are expected to become a major cause of liver disease related deaths and liver transplantation. Currently, there are no specific therapies that alter the natural history of NAFLD.Preliminary evidence suggests that exenatide (Byetta®) may have several beneficial direct and indirect effects on NAFLD and liver lipid metabolism.

DETAILED DESCRIPTION:
Preliminary evidence suggests that exenatide (Byetta®) may have several beneficial direct and indirect effects on NAFLD and liver lipid metabolism. Ad hoc analysis of phase III studies has shown that exenatide treatment is associated with improvement and normalization of alanine aminotransferase (ALT), a marker of liver injury, and that this effect is most pronounced in those with the greatest weight loss. In addition, treatment of leptin deficient ob/ob mice with exenatide reduced weight, liver lipid content, serum ALT and liver lipid peroxidation. Additional evidence suggests that the effects of exenatide on the liver are not simply a result of weight loss, but rather due to direct effects on the liver. Hepatocytes express GLP-1 receptors that are responsive to both GLP-1 and exenatide. Furthermore, exenatide treatment of ob/ob mice or isolated hepatocytes reduces mRNA for stearoyl-CoA desaturase-1 (SCD-1) and SREBP-1c, which would be expected to reduce DNL.

Based upon this data, we hypothesize that exenatide treatment of diabetic patients with NAFLD and NASH will reduce liver injury through multiple mechanisms including weight reduction associated with exenatide, improved lipid metabolism by decreased expression of hepatic genes involved in DNL and reduction of adipokines and cytokines associated with severe NASH. This study is aimed to address the potential safety and efficacy of exenatide in the treatment of NAFLD and test these hypotheses.

This will be an open label, single-arm, non-comparative trial of 20 patients with type 2 diabetes and NAFLD treated with exenatide for 6 months with the following specific aims to be assessed:

Determine the safety and efficacy of 24 weeks of exenatide treatment in diabetic patients with Non-Alcoholic Fatty Liver Disease (NAFLD) Efficacy will be measured by changes in serum ALT (primary endpoint) and liver histology.

Characterize the effects of exenatide on serum levels of adipokines and inflammatory cytokines including adiponectin, leptin and TNF- in NAFLD patients.

Compare the hepatic expression of SCD1, SREBP-1c and PPAR- mRNA in NAFLD patients pre- and post-treatment with exenatide.

Establish the effects of exenatide on post-prandial lipid metabolism.

Determine the effects of exenatide on liver fibrosis in NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, < 70 years, inclusive
* Type 2 diabetes on stable doses of sulfonylurea and/or metformin
* Body mass index > 35 kg/m2
* Presumed diagnosis of NAFLD based upon
* an ALT > 1.5 times the upper limit of reference range,
* no evidence of other causes of liver disease and
* ultrasound findings compatible with fatty liver

Exclusion Criteria:

* Clinical signs of cirrhosis as evidenced by any of the following
* spider angiomata,
* splenomegaly,
* ascites
* jaundice
* encephalopathy
* INR > 1.2
* Platelet count < 100,000/ml
* Serum albumin < 3.0 g/dL
* Other liver disease including chronic viral hepatitis (B or C), alcohol abuse, hemochromatosis, alpha-1 antitrypsin deficiency, autoimmune hepatitis, Wilson's disease, primary sclerosing cholangitis or primary biliary cirrhosis.
* Current use of > 20 g of alcohol per day or unwillingness to avoid alcohol during the course of the study
* Treatment with a thiazolidinedione or exenatide within 6 months of enrolling in the study
* AST or ALT > 10 times the upper limit of normal
* Treatment with any investigational drug within 4 weeks of enrollment
* Pre-menopausal, fertile women unwilling to use contraceptives during the study period.
* Pregnancy or lactation
* Initiation or change in dose of hypolipidemic drugs (statins, niacin, cholestyramine are allowed) within 6 months of enrollment
* Use of anticoagulation, bleeding disorders or other contraindications to liver biopsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Bowlus, MD, Principal Investigator — University of California, Davis; Lars Berglund, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Buse JB, Klonoff DC, Nielsen LL, Guan X, Bowlus CL, Holcombe JH, Maggs DG, Wintle ME. Metabolic effects of two years of exenatide treatment on diabetes, obesity, and hepatic biomarkers in patients with type 2 diabetes: an interim analysis of data from the open-label, uncontrolled extension of three double-blind, placebo-controlled trials. Clin Ther. 2007 Jan;29(1):139-53. doi: 10.1016/j.clinthera.2007.01.015. PMID 17379054
- See also: American Liver Foundation — http://www.liverfoundation.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Alanine aminotransferase [Mean (Full Range); unit: IU] | 84
Glucose [Mean (Full Range); unit: mg/dL] | 139
Cholesterol [Mean (Full Range); unit: mg/dL] | 317
HDL [Mean (Full Range); unit: mg/dL] | 31
Triglyceride [Mean (Full Range); unit: mg/dL] | 482
hsCRP [Mean (Full Range); unit: mg/L] | 8.2
Weight [Mean (Full Range); unit: kg] | 72.3
HbA1c [Mean (Full Range); unit: %] | 8.1

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Serum ALT From Baseline to 24 Weeks of Exenatide Therapy
Time Frame: 24 weeks
Measure: Number; unit: IU
Arm/Group | Exenatide
Number analyzed (Participants) | 1
IU | 61

2. Secondary Outcome: Changes in Components of Liver Histology at Baseline and Week 24 Including Steatosis, Inflammation and Fibrosis
Description: Steatosis was grades on a scale of 0 (< 5%); 1 (5%- 33%); 2 (> 33% - 66%); and 3 (> 66%).
  Inflammation was graded on a scale of 0 (No foci); 1 (< 2 foci per 200 X field); 2 (2-4 foci per 200 X field); and 3 (>4 foci per 200 X field) Fibrosis was graded on a scale of 0 (None); 1 (Mild periportal or perisinusoidal); 2 (Moderate periportal or perisinusoidal); 3 (Bridging fibrosis); and 4 (cirrhosis)
Time Frame: 24 weeks
Measure: Number; unit: units on a scale
Arm/Group | Exenatide
Number analyzed (Participants) | 1
units on a scale
  steatosis | -1
  inflammation | -1
  fibrosis | 0

3. Secondary Outcome: Safety of Exenatide in Patients With NAFLD and Type 2 Diabetes
Time Frame: 24 weeks
Measure: Number; unit: adverse events
Arm/Group | Exenatide
Number analyzed (Participants) | 1
adverse events | 0

ADVERSE EVENTS:
Arm/Group | Exenatide
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No